CLINICAL TRIAL: NCT01264419
Title: SILK ROAD™ MEDICAL EMBOLIC PROTECTION SYSTEM: FIRST IN MAN STUDY "The PROOF Study"
Brief Title: Silk Road Medical First in Man Study - Neuroprotection During Carotid Stenting and Angioplasty
Acronym: PROOF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Silk Road Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRM-2008-01
Record Dates: First submitted 2010-12-17; First posted 2010-12-21 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-01

CONDITIONS: Carotid Artery Diseases
MeSH Terms: conditions — Carotid Artery Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Silk Road Embolic Protection System (Experimental): Eligible subjects who are to receive a carotid artery stent, via transcervical access using reverse flow cerebral protection, as treatment for high-grade extracranial carotid artery disease
  Interventions: Device: Silk Road Embolic Protection System

INTERVENTIONS:
Device: Silk Road Embolic Protection System — System that delivers a carotid artery stent, via transcervical access using reverse flow cerebral protection, as treatment for high-grade extracranial carotid artery disease

SUMMARY:
Cerebral embolization during carotid artery stenting (CAS) can often precipitate severe adverse neurological effects. Most major clinical studies of CAS have used distal filters for cerebral protection and have compared the neurologic complication rates with those of carotid endarterectomy (CEA). Many currently available embolic protection devices, however, have limited efficacy in capturing microembolic debris that is liberated during stenting, pre-dilatation and post-dilatation. Distal protection systems are furthermore limited by the need to cross the lesion prior to deployment. Some studies have shown a relatively high incidence of cerebral infarction even when distal protection devices are employed.

Cerebral protection with carotid flow reversal is a method that was developed by Parodi, et al., as an alternative to the use of distal protection devices. While novel in its approach, this method too has its limitations. Criado, et al., developed a derivative technique that employs carotid flow reversal prior to traversing the stenosis and can be accomplished by directly accessing carotid anatomy without the use of the transfemoral approach. Major benefits to this method include the ability to perform the procedure on patients with severe carotid tortuosity and difficult aortic arch anatomy.

DETAILED DESCRIPTION:
Carotid artery disease is known to increase the risk of neurologic consequences such as transient ischemic attacks (TIA), ischemic stroke, or death due to the release of embolic particles in the vessels supplying the brain. Two principal treatments, carotid endarterectomy (CEA), and carotid artery stenting (CAS), are used to treat this disease. Embolic protection devices, both distal filters and occlusive devices, are employed during the CAS procedure to reduce the risk of carotid plaque embolus secondary to instrumentation during carotid intervention. Existing embolic protection devices are placed using a transfemoral approach and thus have potential for particle embolization while crossing the aortic arch, supraaortic trunk and the carotid lesion before cerebral protection is in place. Other limitations of these devices include the potential for carotid intimal injury, dissection or spasm during deployment, and release of emboli during retrieval.

Noting that carotid embolization remains the "Achilles heel" of carotid artery stenting, an alternative approach to embolic protection was developed by Juan Parodi. The system works by balloon occlusion of the common carotid artery and external carotid artery. An arteriovenous fistula is created with sheaths and catheters and provides retrograde (reverse) blood flow from the internal carotid artery (ICA) and the common carotid artery (CCA) to the femoral vein.

Embolic particles released during CAS pass retrograde through a catheter into a 180 micron filter before the blood re-enters the venous system. (Parodi, Ferreira et al. 2005) A variation of the reverse flow approach utilizing a surgical, transcervical approach to the carotid artery was developed to address challenges and risks associated with the placement and use of existing embolic protection devices. Criado et al. (2004) describe the use of flow reversal during CAS via a transcervical surgical cutdown, access and proximal occlusion of the CCA and establishment of a carotid artery - internal jugular (IJ) vein fistula. (Criado, Doblas et al. 2004).

A difference between the transfemoral-based Parodi approach and the transcervical-based Criado approach is the removal by Criado of the ECA occlusion step. In the Criado approach, the procedure is designed such that the flow is reversed in both the internal and the external carotid arteries, whereas in the Parodi procedure, flow reversal occurs only in the ICA. Another difference in the Criado system is the shorter length and larger diameter tubing afforded by the transcervical approach. The rate of flow reversal enabled by the Criado arteriovenous shunt is higher and is designed to overcome the potential for antegrade flow from the ECA to the ICA.

However, as reported by both Parodi and Criado, active aspiration is often utilized during critical periods of the procedure, to guarantee robust reversal of flow in the ICA.

Similarly in 2004, Chang, et al., reported the use of a direct transcervical approach through a 2cm incision at the base of the neck in 21 CAS patients with a 0% technical failure rate and a 0% thirty-day combined stroke or mortality rate. A similar approach of direct access to the low common carotid artery and the creation of a shunt to the internal jugular was used with carotid occlusion leading to a state of flow reversal. In some cases in this series, a balloon was placed in the external carotid artery. (Chang et al, 2004) Subsequently, Criado et al reported in the Journal of Vascular Surgery in 2004 on a series of fifty patients who underwent carotid artery stenting via this transcervical approach. Using the technique described above, flow was reversed in the ICA by occluding the CCA and establishing a carotid-jugular vein fistula. There was technical success in all 50 procedures and no strokes or deaths occurred. The procedure was tolerated by all but two (4%) of patients. Complications included major and minor carotid artery dissections, which resolved after stent placement. Two transient ischemic attacks (TIA) occurred, one in a patient in whom flow reversal was not successful, and one patient with a contralateral ICA occlusion who suffered a contralateral TIA.(Criado, Doblas et al. 2004).

Criado et al. further report in the Journal of Vascular Surgery in 2004 on a series of 10 awake patients undergoing transcervical carotid artery stenting with flow reversal. Procedural success was achieved in all 10 cases and flow reversal was well tolerated. Cerebral oxygenation during ICA flow reversal was comparable to that during CCA occlusion. ICA angioplasty balloon inflation produced a decrease in SVO2 significantly greater than that occurring during ICA flow reversal. (Criado, Doblas et al. 2004) Finally, Criado et al report on the perioperative and 3 year follow up results of 103 consecutive carotid artery stenting procedures done with a transcervical approach using carotid flow reversal for cerebral protection performed over a 28 month period in 97 patients. Technical success was achieved in 100 cases (97%). No major strokes or deaths occurred. Three awake patients (4%) did not tolerate flow reversal and complications included one ipsilateral TIA, one contralateral TIA, and two minor strokes. There were two wound complications and one major arterial complication. Mean flow reversal time was 21 minutes. At 40 months, the stent patency rate on an intention-to-treat basis was 95%, and the stroke-free survival was 91%. (Criado, Fontcuberta et al. 2007).

In 2006, Ribo and colleagues monitored transcranial doppler (TCD) as part of their standard carotid practice where 23 of 65 patients underwent transcervical carotid stenting using Criado's technique. Mean reversal time was about 15 minutes and well tolerated. TCD monitoring showed an absence of air/solid emboli during stent deployment and angioplasty confirming the presence of reverse flow. Baseline middle cerebral artery (MCA) flow by TCD of 47 cm/sec was substantially decreased with clamping of the common carotid (representing reversal of internal carotid flow). Initial mean antegrade MCA velocity of 30 cm/sec was present post clamping suggesting that there was adequate hemispheric blood flow to be clinically tolerated (Ribo et al. 2006).

Silk Road Medical has developed a system of sheaths, shunts and flow regulators, called the SRM Embolic Protection System, to apply the demonstrated benefits of the Criado and Chang approaches and improve further on ease of use and effectiveness. Silk Road Medical has provided an arteriovenous shunt with the ability to regulate from a low, baseline flow to a higher flow rate. This is accomplished by modulating the flow resistance of a shunt line which connects an arterial and a venous sheath. Because of potential patient intolerance to long periods of high reverse flow, the flow controller enables the user the set the shunt high flow only during periods of the procedure which are high risk for embolic debris (angiography, angioplasty, stent placement). This system eliminates the need for an active aspiration step, and theoretically enables the user to balance patient tolerance needs with optimal embolic protection.

The conclusion from the series of above literature is that transcervical CAS with carotid flow reversal can be accomplished with a high rate of technical success, a very low rate of major adverse events, and an excellent 3 year stroke free survival and stent patency rate. The purpose of this initial investigation is to determine if the SRM Embolic Protection System enables flow reversal of the carotid artery, is compatible with the techniques, devices and equipment used during a carotid artery stenting CAS procedure, and does not present any additional safety risks to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be > 21 years of age.
* Subject has the ability to understand and cooperate with study procedures and agrees to return for all required follow-up visits, tests and exams.
* Subjects taking warfarin may be included if their dosage is reduced before the procedure to result in an International Normalized Ratio (INR) of 1.5 or less. Warfarin may be restarted to therapeutic dose after the procedure.
* The subject must sign a written informed consent prior to the procedure, using a form that is approved by the local medical ethics committee (EC).
* The life expectancy of the subject is at least one year.
* The subject has a lesion located in the internal carotid artery (ICA); the carotid bifurcation may be involved.
* The subject must have a minimum distance of 5 cm between the clavicle and bifurcation, as assessed by duplex Doppler ultrasound, computed axial tomographic (CT) angiography or magnetic resonance (MR) angiography.

Exclusion Criteria:

* The subject was participating in another investigational trial that would interfere with the conduct or result of this study.
* The subject had dementia or a neurological illness that may confound the neurological evaluation.
* Presence of any one of the following anatomic risk factors:

  * Previous radiation treatment to the neck or radical neck dissection
  * Tracheostomy or tracheal stoma
  * Laryngectomy
  * Contralateral laryngeal nerve palsy
  * Severe tandem lesions
  * Inability to extend the head due to cervical arthritis or other cervical disorders
* A total occlusion of the target vessel.
* There was an existing, previously placed stent in the target artery.
* The subject had a known life-threatening allergy to the contrast media that cannot be treated.
* Subject had history of intolerance or allergic reaction to any of the study medications including aspirin, Clopidogrel bisulfate (Plavix®) or Ticlopidine (Ticlid®), heparin or Bivalrudin (Angiomax™). Subject was unable to tolerate a combination of aspirin and Clopidogrel/Ticlopidine.
* The subject had a GI bleed that would interfere with antiplatelet therapy.
* The subject had known cardiac source of potential emboli.
* Subject had a Hemoglobin (Hgb) level less than 8 gm/dL (unless on dialysis), platelet count < 50,000/mm3, or known heparin associated thrombocytopenia.
* Subject had documented atrial fibrillation in the 90 days prior to the procedure.
* The subject had a history of bleeding diathesis or coagulopathy including thrombocytopenia or an inability to receive heparin in amounts sufficient to maintain an Activated Clot Time (ACT) at > 250, or will refuse blood transfusion.
* The subject had atherosclerotic disease involving in the ipsilateral common carotid artery that precluded safe placement of the arterial sheath.
* The subject has other abnormal angiographic findings that indicate the subject is at risk for a stroke due to a problem other than that of the target lesion, such as: ipsilateral arterial stenosis greater in severity than the target lesion, cerebral aneurysm, or arteriovenous malformation of the cerebral vasculature.
* There is evidence of a carotid artery dissection prior to the initiation of the procedure.
* There is an angiographically visible thrombus.
* There is any condition that precludes proper angiographic assessment or makes percutaneous arterial access unsafe, e.g. morbid obesity, sustained systolic blood pressure > 180 mm Hg, tortuosity, occlusive disease, vessel anatomy, aortic arch anatomy, or cerebral protective system.
* Occlusion (TIMI 0 flow), or string sign of the ipsilateral common or internal carotid artery.
* There is evidence of bilateral carotid stenosis that would require intervention within 30 days of procedure.
* There is evidence of a stroke within the previous 30 days of the procedure.
* There is a planned treatment of a non-target lesion within 30 days post procedure.
* There is a history of intracranial hemorrhage within the previous 3 months, including hemorrhagic transformation of an ischemic stroke.
* There is a history of an ipsilateral stroke with fluctuating neurologic symptoms within one year of the procedure.
* Female subjects who are pregnant or may become pregnant.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-03; Primary Completion 2012-06 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sumaira Macdonald, MD, PhD, Study Chair — Chief Medical Officer
Locations (1):
- Augusta-Krankenhaus, Düsseldorf, Germany

REFERENCES:
- [Background] Pinter L, Ribo M, Loh C, Lane B, Roberts T, Chou TM, Kolvenbach RR. Safety and feasibility of a novel transcervical access neuroprotection system for carotid artery stenting in the PROOF Study. J Vasc Surg. 2011 Nov;54(5):1317-23. doi: 10.1016/j.jvs.2011.04.040. Epub 2011 Jun 12. PMID 21658889
- [Result] Alpaslan A, Wintermark M, Pinter L, Macdonald S, Ruedy R, Kolvenbach R. Transcarotid Artery Revascularization With Flow Reversal. J Endovasc Ther. 2017 Apr;24(2):265-270. doi: 10.1177/1526602817693607. Epub 2017 Feb 17. PMID 28335706
- See also: Transcarotid Artery Revascularization With Flow Reversal: The PROOF Study — https://www.ncbi.nlm.nih.gov/pubmed/28335706
- See also: Safety and feasibility of a novel transcervical access neuroprotection system for carotid artery stenting in the PROOF Study. — https://www.ncbi.nlm.nih.gov/pubmed/21658889

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2009 and June 2012 a total of 99 patients were approached about participating in the study. The majority of these individuals (86) were patients of Augusta Krankenhaus in Dusseldorf, Germany, and 13 were patients of the second site, Lukas Krankenhaus, in Neuss, Germany. Study treatment was attempted in 75 study subjects.
Pre-assignment Details: All enrolled participants were assigned to the single arm.
Period: Overall Study
Arm/Group | Silk Road Embolic Protection System
Started | 75
Completed | 72
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- Single: Carotid angioplasty and stenting with Silk Road Embolic Protection System: Major Adverse Event (MAE) rate with reverse flow neuroprotection
Arm/Group | Single
Number analyzed (Participants) | 75
Age, Categorical [Count of Participants; unit: Participants] — Age was reported as such:
  80 years of age or greater; 75 years of age or greater; 70 years of age or greater
  Participants
    <=18 years | 0
    Between 18 and 65 years | 0
    >=65 years | 75
Age, Continuous [Mean (Full Range); unit: years] | 72.61 [70 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety Evaluation as Composite of Occurrences of Major Stroke, Myocardial Infarction and Death
Description: Safety will be evaluated as a composite of major stroke, myocardial infarction and death during the 30-day post procedural period.
Time Frame: 0 days post-procedure to 30 days post-procedure
Population: Per protocol, all enrolled subjects who had a study device placed in their vasculature and completed the 30-day post-procedure period were included in the final analysis data set.
Measure: Number; unit: Occurences
Arm/Group | Silk Road Embolic Protection System
Number analyzed (Participants) | 75
Occurences
  Major Stroke | 0
  Myocardial infarction | 0
  Death | 0

2. Secondary Outcome: Number of Participants Demonstrating Acute Device Success, Procedural Success, and Tolerance to Reverse Flow
Description: Acute Device Success is calculated by tabulating the number of subjects in whom reverse flow could be established AND who received at least 1 stent; Procedural Success is the freedom from MAEs at 30 days post-procedure, where MAEs are defined in the protocol as "A composite rate of death, major stroke, and myocardial infarction (Q wave and non-Q wave)"; Tolerance to Reverse flow is measured as the absence of "any temporary occurrence of procedure related neurological symptoms following the establishment of the cerebral reverse flow circuit that resolves within 20 minutes of flow manipulation". The number of subjects included in "Tolerance to Reverse Flow" were those subjects for whom reverse flow could be both established and measured.
Time Frame: peri-operative to 30 days post-procedure
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Silk Road Embolic Protection System
Number analyzed (Participants) | 75
Participants
  Acute device success | 68
  Procedural Success | 68
  Tolerance to reverse flow: number analyzed (Participants) | 68
  Tolerance to reverse flow | 68

ADVERSE EVENTS:
Arm/Group | Single
Serious Adverse Events (participants affected / at risk) | 10/75
Other Adverse Events (participants affected / at risk) | 48/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single (N=75)
Cranial Nerve Injury (Nervous system disorders) | 2 (2)
Intracranial bleed (Vascular disorders) | 1 (1)
Incorrect Stent Placement (Injury, poisoning and procedural complications) | 1 (1)
Norovirus infection (Gastrointestinal disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
gastrointestinal bleed (Vascular disorders) | 1 (1)
retinopaty associated vision loss (Eye disorders) | 1 (1)
sinus bradycardia (Cardiac disorders) | 1 (1)
Cardiac decompensation with edema (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single (N=75)
Atrial Fibrillation (Cardiac disorders) | 2 (2)
Dyspenia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Procedural vomiting (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 4 (4)
Transient procedure intolerance (Injury, poisoning and procedural complications) | 6 (6)
Vascular access complication (Injury, poisoning and procedural complications) | 4 (4)
Blood potassium decreased (Investigations) | 1 (1)
Full blood count abnormal (Investigations) | 3 (3)
Hemoglobin decreased (Investigations) | 1 (1)
Oxygen Saturation decreased (Investigations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (6)
Sciatica (Nervous system disorders) | 1 (1)
Vertigo (Nervous system disorders) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hematoma (Vascular disorders) | 17 (18)
Hypotension (Vascular disorders) | 5 (5)
Hypertension (Vascular disorders) | 2 (2)
Contact dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Hemorrhage (Vascular disorders) | 3 (3)
Blood CK or CK-MB increase (Investigations) | 3 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Painful Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Tumor excision (Surgical and medical procedures) | 1 (1)
Angina Pectoris (Vascular disorders) | 1 (1)
Cerebral Ischemia (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Standard Non-Disclosure agreement and clinical trial agreement publishing policy in addition.